CLINICAL TRIAL: NCT00885456
Title: Effectiveness of a Program of Rehabilitative Exercise and Education to Avert Vascular Events After Non-disabling Stroke: A Multi-site RCT
Brief Title: Program of Rehabilitative Exercise and Education to Avert Vascular Events After Non-disabling Stroke or Transient Ischemic Attack: A Multi-site RCT
Acronym: PREVENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marilyn MacKay-Lyons (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Stroke Network (Other)
Responsible Party: Sponsor-Investigator, Marilyn MacKay-Lyons, Affiliated Scientist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PREVENT Trial
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Transient Ischemic Attack; Non-disabling Stroke
Keywords: stroke; secondary prevention; vascular risk; behavioral change; exercise; lifestyle modification
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PREVENT program (Experimental): 12-week program of exercise and education to induce physiological and behavioral changes needed to reduce vascular risk factors.
  Interventions: Behavioral: PREVENT program
- Usual Care (Active Comparator): Average of three visits to the Neurovascular Clinic for a neurological and health assessment, counseling regarding stroke/TIA and diagnostic test results, and assessment, modification and education of secondary prevention factors
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: PREVENT program — 12-week program of aerobic/strengthening exercises and education designed to induce physiological and behavioral changes deemed necessary to reduce vascular risk
  Arms: PREVENT program
Behavioral: Usual Care — Three or more out-patient visits to the neurovascular clinic for assessment, counseling and referral to appropriate health care professionals.
  Arms: Usual Care

SUMMARY:
The objective of the Program of Rehabilitative Exercise and Education to avert Vascular Events after Non-disabling stroke and Transient ischemic attack (PREVENT) Trial is to determine whether the timely delivery of secondary stroke prevention strategies will reduce modifiable vascular risk factors in two groups of people who have survived NDS or TIA. One group will receive a comprehensive education and exercise program (PREVENT); the other group will receive usual care (USUAL CARE). We will measure modifiable vascular risk factors in both groups. We will also compare the effects of PREVENT vs USUAL CARE on exercise capacity, walking endurance, and daily physical activity. In addition, we will compare thinking ability, depression, achievement of personal goals for healthy behavior, and health-related goal attainment and health-related quality of life. Finally, we will compare outcomes in urban and rural settings as well as costs of the PREVENT program and USUAL CARE in order to assess sustainability of the PREVENT program.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Over 17 years of age.
* Diagnosis of first probable or definite TIA or non-disabling stroke (National Institutes of Health Stroke Scale < 6)
* Post-event interval of <90 days.
* Residence within 75 km of intervention site.
* Orientation to time, place and person and ability to follow simple 3-step commands.
* Ability and willingness to provide informed consent.

Exclusion Criteria:

* Evidence of intracranial hemorrhage on MRI or CT scan.
* Presence of contraindications to exercise testing and training, in accordance with American College of Sports Medicine Guidelines.
* Participation in another study that could potentially confound the outcomes of this trial.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2011-10-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure (primary vascular risk factor being assessed) | baseline, post-intervention, 6 months, 12 months
diastolic blood pressure | baseline, post-intervention, 6 months, 12 months
waist circumference | baseline, post-intervention, 6 months, 12 months
12-hour fasting lipid profile | baseline, post-intervention, 6 months, 12 months
12-hour fasting glucose/hemoglobin A1C | baseline, post-intervention, 6 months, 12 months

SECONDARY OUTCOMES:
exercise capacity | baseline, post-intervention, 12 months
daily physical activity | baseline, post-intervention, 6 months, 12 months
walking endurance | baseline, post-intervention, 6 months, 12 months
cigarette smoking | baseline, post-intervention, 6 months, 12 months
medication adherence | baseline, post-intervention, 6 months, 12 months
cognition | baseline, 12 months
depression | baseline, post-intervention, 6 months, 12 months
health-related quality of life | baseline, post-intervention, 6 months, 12 months
health-related goal attainment | baseline, post-intervention, 6 months, 12 months
direct health costs | baseline, post-intervention, 6 months, 12 months
secondary vascular events | baseline, post-intervention, 6 months, 12 months
daily step count | baseline, post-intervention, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn MacKay-Lyons, PhD, Principal Investigator — Dalhousie University
Locations (2):
- Canada (2):
  - Halifax Infirmary Site, QEII Health Sciences Centre, Halifax, Nova Scotia
  - Annapolis Valley Regional Hospital, Kentville, Nova Scotia

REFERENCES:
- [Derived] MacKay-Lyons M, Gubitz G, Phillips S, Giacomantonio N, Firth W, Thompson K, Theriault C, Wightman H, Slipp S, Marsters D, Eskes G, Peacock F, Blanchard C, Dewolfe J. Program of Rehabilitative Exercise and Education to Avert Vascular Events After Non-Disabling Stroke or Transient Ischemic Attack (PREVENT Trial): A Randomized Controlled Trial. Neurorehabil Neural Repair. 2022 Feb;36(2):119-130. doi: 10.1177/15459683211060345. Epub 2021 Nov 17. PMID 34788569
- [Derived] MacKay-Lyons M, Gubitz G, Giacomantonio N, Wightman H, Marsters D, Thompson K, Blanchard C, Eskes G, Thornton M. Program of rehabilitative exercise and education to avert vascular events after non-disabling stroke or transient ischemic attack (PREVENT Trial): a multi-centred, randomised controlled trial. BMC Neurol. 2010 Dec 8;10:122. doi: 10.1186/1471-2377-10-122. PMID 21143864